CLINICAL TRIAL: NCT01588353
Title: Phase III Study of AK160 in Patients With Dupuytren's Contracture
Brief Title: Collagenase Option for Reduction of Dupuytren's Contracture in Japan
Acronym: CORD-J
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK160-III-1
Record Dates: First submitted 2012-04-27; First posted 2012-04-30 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Dupuytren's Contracture
Keywords: AK160, collagenase clostridium histolyticum
MeSH Terms: conditions — Dupuytren Contracture | interventions — Microbial Collagenase; xiapex

ARMS (1):
- AK160 0.58 mg (Experimental)
  Interventions: Drug: Collagenase Clostridium Histolyticum

INTERVENTIONS:
Drug: Collagenase Clostridium Histolyticum — AK160 (Collagenase Clostridium Histolyticum) 0.58 mg
  Other Names: Xiaflex® (US); Xiapex® (EU)

SUMMARY:
To investigate the efficacy and safety of AK160 in patients with Dupuytren's Contracture.

To determine plasma concentration after the first injection of AK160 in patients with Dupuytren's Contracture.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years old when written informed consent is obtained.
* Having a diagnosis of Dupuytren's contracture and flexion contracture due to palpable cord in at least 1 non-thumb finger (20° to 100° in MP joint and 20° to 80° in PIP joint).
* Positive tabletop test result (i.e., cannot simultaneously place affected finger and palm on a table).
* Voluntary written informed consent is obtained.

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded:

* Is pregnant, may be pregnant, wishes to become or could become pregnant during the study (i.e., unless acceptable contraception is used, the patient has been sterilized, or the patient is postmenopausal [no menstrual period for at least 12 months without any other medical cause]), or is breastfeeding.
* Has a coexisting chronic disease of the hand that could impact assessment (muscular disease, neurological disease, neuromuscular disease).
* Has received another investigational product 30 or fewer days before first injection of the investigational product.
* Has undergone aponeurectomy, aponeurotomy, needle aponeurotomy/fasciotomy, verapamil/interferon injection, or another Dupuytren's Contracture treatment of the primary joint 90 or fewer days before first injection of the investigational product.
* Is allergic to collagenase or any of the excipients of AK160.
* Has taken tetracycline derivative such as minocycline and doxycycline 14 or fewer days before first injection of the investigational product.
* Has received a collagenase product 30 or fewer days before first injection of the investigational product.
* Is currently taking or has taken, 7 or fewer days before first injection of the investigational product, an anticoagulant or antiplatelet drug (other than ≤150 mg/day of aspirin).
* Has suffered a recent stroke, hemorrhage, or other disease affecting the hands.
* Has a serious disease unsuited for the study.
* Receiving treatment for a malignancy.
* History of drug or alcohol addiction within the past 5 years or history of drug or alcohol abuse within the past year.
* Has received previously the investigational product (AK160, AA4500, XIAFLEX®, or XIAPEX®).
* Otherwise found ineligible as a subject by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- Japan (20):
  - Aichi
  - Aomori
  - Chiba
  - Fukuoka
  - Hiroshima
  - Hokkaido
  - Ishikawa
  - Kanagawa
  - Kumamoto
  - Kyoto
  - Mie
  - Nagano
  - Nagasaki
  - Niigata
  - Numakunai
  - Okayama
  - Osaka
  - Tokushima
  - Tokyo
  - Yamaguchi

REFERENCES:
- [Result] Hirata H, Tanaka K, Sakai A, Kakinoki R, Ikegami H, Tateishi N. Efficacy and safety of collagenase Clostridium histolyticum injection for Dupuytren's contracture in non-Caucasian Japanese patients (CORD-J Study): the first clinical trial in a non-Caucasian population. J Hand Surg Eur Vol. 2017 Jan;42(1):30-38. doi: 10.1177/1753193416653249. Epub 2016 Sep 28. PMID 27313184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 104 patients were enrolled, and 102 received AK160. This study proceeded stepwise from Step1 through Step3. First, 6 patients were enrolled in Step1 at the selected study centers, thereafter, 71 and 25 patients were enrolled in Steps2 and3 respectively at all centers. The primary endpoint was determined in 77 participants enrolled in Steps1 and 2.
Groups:
- AK160 0.58 mg Step1: This arm consisting of participants enrolled in step 1 was used to confirm the efficacy and satety of the drug 30 days after the first dose before starting step 2.
  And also this arm was used to determine the efficacy of the drug with participants enrolled in step 2 and to determine the safety with participants enrolled in steps 2 and 3.
  Collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal(PIP) joints. Collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints.
- AK160 0.58 mg Step 2: This arm consisting of participants enrolled in step 2 was used to determine the efficacy of the drug with participants enrolled in step 1 and to determine the safety with participants enrolled in steps 1 and 3.
  Collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal(PIP) joints. Collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints.
- AK160 0.58 mg Step3: The participants in step 3 were added until the number of injected joints by joint type became up to 50 or more in steps1 through 3.
  This arm was mainly used to determine the safety of the drug with participants enrolled in steps 1 and 2.
  Collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal(PIP) joints. Collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints.
Period: Step1
Arm/Group | AK160 0.58 mg Step1 | AK160 0.58 mg Step 2 | AK160 0.58 mg Step3
Started | 6 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Step2
Arm/Group | AK160 0.58 mg Step1 | AK160 0.58 mg Step 2 | AK160 0.58 mg Step3
Started | 0 | 71 | 0
Completed | 0 | 70 | 0
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Step3
Arm/Group | AK160 0.58 mg Step1 | AK160 0.58 mg Step 2 | AK160 0.58 mg Step3
Started | 0 | 0 | 25
Completed | 0 | 0 | 23
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- AK160 0.58 mg Step 1: This arm consisting of participants enrolled in step 1 was used to confirm the efficacy and satety of the drug 30 days after the first dose before starting step 2.
  And also this arm was used to determine the efficacy of the drug with participants enrolled in step 2 and to determine the safety with participants enrolled in steps 2 and 3.
  Collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal(PIP) joints. Collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints.
- Total: Total of all reporting groups
Arm/Group | AK160 0.58 mg Step 1 | AK160 0.58 mg Step 2 | AK160 0.58 mg Step3 | Total
Number analyzed (Participants) | 6 | 71 | 25 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 22 | 2 | 26
  >=65 years | 4 | 49 | 23 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (8.3) | 68 (8.4) | 71 (5.9) | 68.7 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 3 | 10
  Male | 5 | 65 | 22 | 92
Region of Enrollment [Number; unit: participants]
  Japan | 6 | 71 | 25 | 102

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants That Were Successfully Treated With a "Successful Reduction in Contracture to 5°or Less"
Description: The Primary Outcome Measure for participants who were enrolled at Step1 through Step2 and treated with AK160 is the percentage of 77 participants that were successfully treated where "successfully treated" was defined as reduction in the contracture of the first treated joint to 5° or less. The injection was allowed up to 3 times.
Time Frame: 30 days after the last injection
Population: The primary efficacy analysis population was the full analysis set (FAS) comprising subjects treated with study drug in Steps 1 and 2.
Measure: Number; unit: % Participants
Groups:
- AK160 0.58 mg Step 1-2: collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints
Arm/Group | AK160 0.58 mg Step 1-2
Number analyzed (Participants) | 77
% Participants | 86

2. Secondary Outcome: Clinical Improvement After the Last Injection
Description: The Secondary Outcome Measure for participants who were enrolled at Step1 through Step2 and treated with AK160 is the percentage of 77 participants that were clinically improved where "clinically improved" was defined as reduction in the contracture of the first treated joint by 50% or more from the baseline. The injection was allowed up to 3 times.
Time Frame: 30 days after the last injection
Population: The secondary efficacy analysis population was the full analysis set (FAS) comprising subjects treated with study drug in Steps 1 and 2.
Measure: Number (95% Confidence Interval); unit: % Participants
Groups:
- Primary MP Joints: collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) joints
- Primary PIP Joints: collagenase clostridium histolyticum 0.58mg injected into proximal interphalangeal (PIP) joints
- Total: collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) or proximal interphalangeal (PIP) joints
Arm/Group | Primary MP Joints | Primary PIP Joints | Total
Number analyzed (Participants) | 47 | 30 | 77
% Participants | 100 [92.5 to 100.0] | 90.0 [73.5 to 97.9] | 96.1 [89.0 to 99.2]

3. Secondary Outcome: Percent Reduction From Baseline Contracture After the Last Injection
Description: The Secondary Outcome Measure for participants who were enrolled at Step1 through Step2 and treated with AK160 is the mean percent decrease from baseline degree of contracture in primary joints after the last injection. The injection was allowed up to 3 times.
Time Frame: 30 days after last treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of change from baseline
Arm/Group | Primary MP Joints | Primary PIP Joints | Total
Number analyzed (Participants) | 47 | 30 | 77
% of change from baseline | 97.08 (7.791) | 82.48 (24.674) | 91.39 (17.900)

4. Secondary Outcome: Change From Baseline Range of Motion After the Last Injection
Description: The Secondary Outcome Measure for participants who were enrolled at Step1 through Step2 and treated with AK160 is the change from baseline range of motion in primary joints after the last injection. The injection was allowed up to 3 times.
Time Frame: 30 days after last treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Primary MP Joints | Primary PIP Joints | Total
Number analyzed (Participants) | 47 | 30 | 77
Degrees | 41.6 (18.91) | 33.3 (17.73) | 38.4 (18.79)

5. Secondary Outcome: Time to First Achieve and Maintain Clinical Success After the Last Injection
Description: The Secondary Outcome Measure for participants who were enrolled at Step1 through Step2 and treated with AK160 is the time to first achieve and maintain clinical success after the last injection where "clinical success" was defined as reduction in the contracture of the first treated joint to 5° or less. The injection was allowed up to 3 times.
Time Frame: First evaluation visit on which clinical success is achieved and maintained through the Day 30 evaluation of each injections, assessed up to 3 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Primary MP Joints | Primary PIP Joints | Total
Number analyzed (Participants) | 47 | 30 | 77
Days | 1.0 [1.0 to 28.0] | 7.0 [1.0 to 92.0] | 1.0 [1.0 to 30.0]

ADVERSE EVENTS:
Time Frame: Adverse events were investigated from the day of the first injection of the study drug until 360 days after the first injection of the study drug.
Groups:
- AK160 0.58 mg Step 1-3: Collagenase Clostridium Histolyticum: AK160 (Collagenase Clostridium Histolyticum) 0.58 mg
Arm/Group | AK160 0.58 mg Step 1-3
Serious Adverse Events (participants affected / at risk) | 14/102
Other Adverse Events (participants affected / at risk) | 100/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AK160 0.58 mg Step 1-3 (N=102)
Cataract (Eye disorders) | 3 — All were determined by investigators to be not related to the study drug.
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — All were determined by investigators to be not related to the study drug.
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — All were determined by investigators to be not related to the study drug.
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — All were determined by investigators to be not related to the study drug.
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 — All were determined by investigators to be not related to the study drug.
Intestinal obstruction (Gastrointestinal disorders) | 1 — All were determined by investigators to be not related to the study drug.
Infectious pleural effusion (Infections and infestations) | 1 — All were determined by investigators to be not related to the study drug.
Bile duct stone (Hepatobiliary disorders) | 1 — All were determined by investigators to be not related to the study drug.
Spondylolysis (Musculoskeletal and connective tissue disorders) | 1 — All were determined by investigators to be not related to the study drug.
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 — All were determined by investigators to be not related to the study drug.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 — All were determined by investigators to be not related to the study drug.
Myocardial infarction (Cardiac disorders) | 1 — All were determined by investigators to be not related to the study drug.
Subarachnoid haemorrhage (Nervous system disorders) | 1 — All were determined by investigators to be not related to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AK160 0.58 mg Step 1-3 (N=102)
Injection site pain (General disorders) | 78
Injection site bruising (General disorders) | 46
Injection site swelling (General disorders) | 35
Contusion (Injury, poisoning and procedural complications) | 30
Injection site laceration (General disorders) | 16
Nasopharyngitis (Infections and infestations) | 16
Injection site oedema (General disorders) | 12
Injection site haematoma (General disorders) | 11
Local swelling (General disorders) | 9
Laceration (Injury, poisoning and procedural complications) | 9
Lymphadenitis (Blood and lymphatic system disorders) | 6
Injection site pruritus (General disorders) | 6
Glucose urine present (Investigations) | 6
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Asahi Kasei Pharma Corporation agreements may vary with individual facilities but will not prohibit any investigator from publishing. Asahikasei supports the publication of results from all centers of a multicenter trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.